CLINICAL TRIAL: NCT06555965
Title: STXBP1 and SYNGAP1 Related Disorders (RD) Natural History Study
Brief Title: STXBP1 and SYNGAP1 Related Disorders Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: STXBP1 Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23-021140
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Genetic Disease; STXBP1 Encephalopathy With Epilepsy; SYNGAP1-Related Intellectual Disability
Keywords: STXBP1; Natural History; Clinical Research; SYNGAP1
MeSH Terms: conditions — Genetic Diseases, Inborn; Epileptic Encephalopathy, Early Infantile, 4

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STXBP1 cohort
  Interventions: Other: Non-interventional study
- SYNGAP1 cohort
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — There is no planned intervention in this study

SUMMARY:
The purpose of this study is to find out more about STXBP1 and SYNGAP1 related disorders. The information gathered by this study will be used to prepare for clinical treatment trials. The primary objective of the study is to better define and outline the clinical spectrum of STXBP1 and SYNGAP1 through detailed developmental, seizure, and quality of life assessments as an extension of routine clinical care.

DETAILED DESCRIPTION:
STXBP1 and SYNGAP1 related disorders are genetic disorders that cause differences in the synaptic transmission of the brain. Disease-causing variants in these genes lead to a spectrum of developmental delay that is most often severe, epileptic encephalopathies, and complex behavioral and psychiatric disorders. As there are multiple targeted therapies in development for these conditions, there is an urgent need to push forward a prospective natural history study in order to define specific disease outcomes in these genetic conditions.

Participation may last up to five years and will involve up to 10 study visits. Detailed questions about health and medical history, physical exams, electrographic encephalogram (EEG) or quantitative EEG (qEEG) and some age-appropriate assessments of neurodevelopmental and behavioral function are some of the study procedures. Study procedures will occur during regularly scheduled clinic visits. Participants will undergo assessments at baseline visit and semi-annually (every 6 months for 2-5 years).

The primary objective of the study is to better define and outline the clinical spectrum of STXBP1 and SYNGAP1 through detailed developmental, seizure, and quality of life assessments as an extension of routine clinical care.

The secondary objectives of the study are listed below:

* To evaluate changes in neurodevelopmental and behavioral parameters as assessed by instruments appropriate to the study population.
* To assess the burden of disease by quality-of-life instruments appropriate to the study population.
* To assess the burden of performing multiple outcome measures and scales on the caregiver, participant, and clinical personnel.
* To assess health care resource utilization

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age.
* Presence of a STXBP1 or SYNGAP1 gene mutation. The variant in STXBP1 or SYNGAP1 must be classified as causative based on clinical and variant classification criteria. Historical documentation is sufficient to support eligibility for the study. Confirmatory testing will be obtained, if necessary, at baseline and performed by a CLIA certified laboratory.

Exclusion Criteria:

* The presence of a confirmed mutation in a gene other than STXBP1 or SYNGAP1 that is known to contribute to a neurodevelopmental disability. This includes full gene deletions of STXBP1 or SYNGAP1 that include other genes beyond STXBP1 or SYNGAP1.
* The presence of a significant non-STXBP1-RD or non-SYNGAP1-RD related central nervous impairment/behavioral disturbance that would confound the scientific rigor or interpretation of results of the study.
* History of intraventricular hemorrhage, structural brain deficit or congenital heart disease
* The presence of a clinical comorbidity deemed by the investigator to potentially confound the typical presentation of STXBP1-RD or SYNGAP1-RD.
* Pregnant women or females of age of menarche who are found to be pregnant upon urine pregnancy testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participating individuals must have a confirmed genetic diagnosis of STXBP1 or SYNGAP1 related disorders. Participants can be any age and present with any disease severity
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2028-08-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in percentiles recorded on clinical assessments over time | Every 6 months upto 5 years
  The primary analysis will include all subjects meeting all inclusion and exclusion criteria and completing Visit 1. For each subject, the percentage of items performed correctly on the clinical assessments will be recorded. Changes in percentiles over time will be analyzed using a linear mixed effects model, to account for repeated measures for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Helbig, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Stanford Medicine Children's Health, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Weill Cornell Medicine, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xian J, Parthasarathy S, Ruggiero SM, Balagura G, Fitch E, Helbig K, Gan J, Ganesan S, Kaufman MC, Ellis CA, Lewis-Smith D, Galer P, Cunningham K, O'Brien M, Cosico M, Baker K, Darling A, Veiga de Goes F, El Achkar CM, Doering JH, Furia F, Garcia-Cazorla A, Gardella E, Geertjens L, Klein C, Kolesnik-Taylor A, Lammertse H, Lee J, Mackie A, Misra-Isrie M, Olson H, Sexton E, Sheidley B, Smith L, Sotero L, Stamberger H, Syrbe S, Thalwitzer KM, van Berkel A, van Haelst M, Yuskaitis C, Weckhuysen S, Prosser B, Son Rigby C, Demarest S, Pierce S, Zhang Y, Moller RS, Bruining H, Poduri A, Zara F, Verhage M, Striano P, Helbig I. Assessing the landscape of STXBP1-related disorders in 534 individuals. Brain. 2022 Jun 3;145(5):1668-1683. doi: 10.1093/brain/awab327. PMID 35190816
- [Background] Yang P, Broadbent R, Prasad C, Levin S, Goobie S, Knoll JH, Prasad AN. De novo STXBP1 Mutations in Two Patients With Developmental Delay With or Without Epileptic Seizures. Front Neurol. 2021 Dec 24;12:804078. doi: 10.3389/fneur.2021.804078. eCollection 2021. PMID 35002943
- [Background] Wang HH, Liao HF, Hsieh CL. Reliability, sensitivity to change, and responsiveness of the peabody developmental motor scales-second edition for children with cerebral palsy. Phys Ther. 2006 Oct;86(10):1351-9. doi: 10.2522/ptj.20050259. PMID 17012639
- [Background] Demarest S, Pestana-Knight EM, Olson HE, Downs J, Marsh ED, Kaufmann WE, Partridge CA, Leonard H, Gwadry-Sridhar F, Frame KE, Cross JH, Chin RFM, Parikh S, Panzer A, Weisenberg J, Utley K, Jaksha A, Amin S, Khwaja O, Devinsky O, Neul JL, Percy AK, Benke TA. Severity Assessment in CDKL5 Deficiency Disorder. Pediatr Neurol. 2019 Aug;97:38-42. doi: 10.1016/j.pediatrneurol.2019.03.017. Epub 2019 Mar 27. PMID 31147226